CLINICAL TRIAL: NCT01150812
Title: A Phase I, Single-center, Single-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD8165 After Single Oral Ascending Doses in Healthy Male Subjects
Brief Title: Oral AZD8165 After Single Oral Ascending Doses in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study pharmacodynamic stopping criteria were met after the first dosing group
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D2890C00001
Record Dates: First submitted 2010-06-21; First posted 2010-06-25 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Thrombin Inhibition
Keywords: First time in man; healthy; thrombin inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD8165

INTERVENTIONS:
Drug: AZD8165 — Oral suspension, 2 mg/mL and 20 mg/mL, single doses

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of AZD8165 and the pharmacokinetics of the metabolite AZ12971554 and plasma levels of the prodrug AZD8165 after escalating single oral low doses.

ELIGIBILITY:
Inclusion Criteria:

* Suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and nor more than 100 kg

Exclusion Criteria:

* History of any clinically significancy disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Personal or family history of bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, Electrocardiograms, vital signs, safety labs) | Approximately 64 days including a screening period, 3 treatment periods, 2 washout periods, and a follow-up period.

SECONDARY OUTCOMES:
Plasma and urine levels of AZD8165 and its active metabolite AZ12971554 | Serial blood and urine samples will be taken over 24 hours after oral administration to evaluate AZD8165 and its active metabolite AZ12971554
Coagulation times (namely Activated Partial Thromboplastin Time,Ecarin Clotting Time, Thrombin Clotting Time | Serial blood samples will be taken over 24 hours after oral administration to evaluate Activated Partial Thromboplastin Time (APTT), Ecarin clotting Time (ECT), Thrombin Clotting Time (TCT)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schutz, MD, Principal Investigator — Quintiles, Inc.; Peter Held, Study Director — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States